CLINICAL TRIAL: NCT02789215
Title: Proposed Meal Changes for CACFP: Impact on Child Food Intake and Costs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jayna Dave, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-35784; R01HL119520 (NIH)
Record Dates: First submitted 2016-05-25; First posted 2016-06-02 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Food Security
Keywords: Child care food costs; Meal participation rates; Child and Adult Care Food Program
MeSH Terms: interventions — Costs and Cost Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Receive new CACFP menu pattern
  Interventions: Behavioral: Proposed Meal Changes for CACFP: Impact on Child Food Intake and Costs
- Control (No Intervention): Follow existing CACFP menu pattern

INTERVENTIONS:
Behavioral: Proposed Meal Changes for CACFP: Impact on Child Food Intake and Costs
  Arms: Intervention

SUMMARY:
Child and Adult Care Food Program (CACFP) meals are an important influence on diets of children from low-income families enrolled in the CACFP and should meet children's nutrient needs while fostering healthy eating habits that enable them to maintain energy balance. Recent national data revealed that children consumed low intakes of foods that support healthy dietary patterns (whole grains, fruit and vegetables other than potatoes), but high intakes of low nutrient, energy dense foods. The 2011 USDA-commissioned Institute of Medicine (IOM) report for CACFP meals provided new recommendations that include new meal pattern requirements for the meals programs, aligning them with the U.S. Dietary Guidelines to ensure that the meals promote health and reduce inadequate and excessive intakes. The report recommended inclusion of more whole grains, fruit, vegetables, and meat/meat alternatives which will likely increase meal costs. Two of the IOM report recommendations call for research to better understand how the new meal requirements would change children's CACFP meal dietary intakes and food service costs. These are important questions, and answers are needed to inform policy and future technical and educational assistance needs. The overall objective of this project is to implement the IOM meal pattern requirements for CACFP meals in day homes and centers in Texas. The multidisciplinary team will focus on nutrition, economics, and provider outcomes. The specific aims are to assess the impact of the new meal pattern requirements on 1) Meal participation rates; 2) Provider food service costs (food, labor, total meals); and 3) Child dietary intake at CACFP homes and centers. It is hypothesized that, compared with control sites, intervention site children will select and consume healthier diets (more fruit, vegetables and whole grains) at school. A total of 32 day care sites will be recruited for the study. It is hypothesized that, compared with control sites, children at the intervention sites will select and consume healthier diets (more fruit, vegetable and whole grains) at the center. It is also hypothesized that the increase in food costs will be less than that projected in the IOM report. The results on the costs associated with creating the desired meals will be very important as these data have not been systematically collected in previous studies. This significant study targets underserved minority populations with health promoting intervention to reduce health disparities, and in addition, will inform policy on the influence of a healthy food environment on children's diet, as well as provide critical information on costs.

ELIGIBILITY:
Inclusion Criteria:

* Must be day care sites
* Must be parents of children attending the day care sites

Exclusion:

* Parents of children not attending one of the 32 day care sites

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Child Dietary Intake at 6 months and 12 months | Up to 12 months
Change from Baseline Meal Participation Rates at 6 months and 12 months | Up to 12 months
Change from Baseline Provider Food Service Costs (food, labor, total meals) at 6 months and 12 months | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The Baylor College of Medicine understands and agrees to comply with the NIH policy on Sharing Research Data and on Sharing Model Organisms (as outlined in the NIH Guide, February 26, 2003 and May 7, 2004.) The principal investigator and co-investigators acknowledge their willingness to share data and materials with other eligible investigators through academically established means. Data will be shared with collaborators as soon as available, with local colleagues at seminars and talks, and with the scientific community at large by posters and presentations at local, regional, national and international scientific meetings. Finally, data will be presented by publication to the widest audience possible. Press interviews on important publications are arranged through the Baylor College of Medicine Office of Public Affairs.

REFERENCES:
- [Result] Dave JM, Cullen KW. Foods Served in Child Care Facilities Participating in the Child and Adult Care Food Program: Menu Match and Agreement with the New Meal Patterns and Best Practices. J Nutr Educ Behav. 2018 Jun;50(6):582-588. doi: 10.1016/j.jneb.2018.01.010. Epub 2018 Feb 21. PMID 29475767
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/29475767